CLINICAL TRIAL: NCT02659527
Title: Randomized Assessment of Patients With Clinically Suspected Prostate Cancer After Multiparametric Metabolic Hybrid Imaging to Evaluate Its Potential Clinical Domain: A Prospective, Randomized, Multi-arm, Multi-treatment Clinical Trial
Brief Title: PET/MRI in Patients With Suspected Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: BSM Diagnostica GmbH Vienna (Unknown); Siemens Healthcare GmbH (Unknown)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Marcus Hacker, Univ.-Prof. Dr.med, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: The RAPID study
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standardized needle biopsy (Active Comparator): All enrolled patients are examined by means of dual tracer PET / MRI. Images will be interpreted by 4 designated readers. The readers are blinded of the respective results among each other. A consensus of the two principal readers of nuclear medicine and radiology will serve as reference for the guided needle biopsy. Additionally the readers are blinded to any result of the pathological workout until the recruitment of the last patient is finished.
  According to the randomization, the standardized 12 core TRUS (TransRectal UltraSound)-guided biopsy is performed without knowledge of imaging findings by the urologist. If the biopsy is negative patients will have an additional image-guided biopsy with 4 more cores samples. After a positive biopsy the subjects be treated according to normal clinical practice.
  Interventions: Drug: 68Ga- PSMA-HBED-CC; Device: Biograph mMR, Siemens
- image-guided biopsy (Experimental): All enrolled patients are examined by means of dual tracer PET / MRI. Images will be interpreted by 4 designated readers. The readers are blinded of the respective results among each other. A consensus of the two principal readers of nuclear medicine and radiology will serve as reference for the guided needle biopsy. Additionally the readers are blinded to any result of the pathological workout until the recruitment of the last patient is finished.
  Patients will have a standardized 12 core TRUS-guided biopsy without knowledge of imaging findings by the urologist. Patients randomized in this arm will have an additional image-guided biopsy with 4 more cores samples. After a positive biopsy the subjects be treated according to normal clinical practice.
  Interventions: Drug: 68Ga- PSMA-HBED-CC; Device: Biograph mMR, Siemens

INTERVENTIONS:
Drug: 68Ga- PSMA-HBED-CC — Patients will receive a dual-tracer PET/MRI scan. FEC and 68Ga-PSMA-HBED-CC, for tissue metabolism and surface marker expressions, as specific PET-tracers as well as multiparametric MRI methods (T2w, DCE, DWI) are used.
Device: Biograph mMR, Siemens — All PET-MRI examinations will be performed using a hybrid PET-MRI system (Biograph mMR, Siemens, Germany) capable of simultaneous data acquisition. The system consists of an MRI-compatible state-of the art PET detector integrated in a 3.0-T whole-body MRI scanner.

SUMMARY:
This diagnostic clinical trial will be conducted according to a randomized, prospective, controlled, double-arm, single-centre design. The control will be implemented by comparing the PET/MRI results with the histopathological finding after radical prostatectomy (positive state), the assumed absence of a relevant prostate cancer focus if PET/MRI guided biopsy and standard biopsy are negative (negative state) and/or the detection of a biochemical tumor relapse [rising prostate specific antigen (PSA) after PSA nadir; secondary objective].

DETAILED DESCRIPTION:
In the last years magnetic resonance imaging (MRI) as well as positron emission tomography (PET) of the prostate have emerged as promising imaging tools. MRI provides mainly morphologic information and, to an increasing degree, functional information on the tumor microenvironment by using multiparametric approaches leading to an increase in diagnostic accuracy. Transition and periurethral zone cancers and the identification of patients' individual risk (e.g. for the development of a metastatic disease after primary treatment) is still a limitation of this method. PET, concerning radiolabelled choline, provides functional and predicting data on tumor metabolism and aggressiveness and has been found to be of complimentary value to morphologic imaging but still with the caveat of false positive and false negative findings. To overcome these limitations of morphological and functional imaging techniques, hybrid imaging systems have been developed and introduced into clinical routine. Additionally, the recently developed 68Ga-labeled Prostate Specific Membrane Antigen (PSMA) provides a highly specific information on a possible metastatic spread of prostate cancer. Thus the combined use of PET-MRI has wide spread applications in prostate cancer diagnosis, staging and treatment planning.

The potentials of this novel technique in general and its impact on assessing patients' individual risk to support a therapy or active surveillance decision in a future modified urological patient management were not yet explored in detail, but an initial prospective clinical trial in 38 patients with a sequential PET/MRI technique demonstrated the ability of a significant improvement of the individual methods. This registered prospective, randomized clinical trial is intended to proof, in a first step, the superiority of PET/MRI vs. the actual clinical standard procedures by applying a stable multiparametric metabolic hybrid imaging protocol. The aim of this study is to reduce the number of unnecessary invasive procedures to a minimum (image guided biopsy) and to enable superior image guided risk stratification.

In this prospective, randomized, multi-arm, multi-treatment clinical trial 220 subjects will be included at 1 site within 3 years. With a maximum follow-up for an early biochemical relapse of 2 years the planned duration should not exceed 5 years. The primary objective will be answered after 36 months.

ELIGIBILITY:
Inclusion Criteria:

* blood PSA level > 4.0 ng/ml and
* free-to-total PSA ratio <22% and/or
* progressive rise of PSA levels in two consecutive blood samples despite antibiotics

Exclusion Criteria:

* antiandrogen therapy
* prostate needle biopsy <21 days before PET/MRI
* known active secondary cancer
* endorectal coil not applicable (e.g. anus praetor with short rectal stump)
* known active prostatitis (e.g. painful DRE)
* known anaphylaxis against gadolinium-DOTA
* patient's written informed consent not given
* needle biopsy and/or prostatectomy compound not available for histology/immunohistochemistry

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Superiority of image guided biopsy using multiparametric metabolic hybrid imaging with FEC/PSMA-PET/MRI (Fluorethylcholin/Prostate Specific Membrane Antigen- PET/MRI) | 36 months
  We hypothesize that the image guided biopsy using multiparametric metabolic hybrid imaging with FEC/PSMA-PET/MRI is superior in the detection of primary localized prostate cancer than the conventional biopsy approach with transrectal ultrasound in patients with suspected prostate cancer (according to the inclusion criteria) and could therefore significantly improve the detection rate of the dominant intraprostatic tumor lesion and reduce the number of biopsies needed for a correct histopathological diagnosis to a minimum in the future (PET/MRI guided biopsy).

SECONDARY OUTCOMES:
tumor characterization | 5 years
  This method should enable improved tumor characterization. A diagnostic accuracy of >80% is assumed in lesions >5mm (in axial, sagittal and coronal extension) for the ability of the multiparametric metabolic method to differentiate between Gleason ≤3+4=7 (7a) tumors and ≥4+3=7 (7b) tumors (as compared to histological whole mount tumor mapping) and to identify patients with a high risk of developing metastatic disease (as compared to the loss of the transcription factor STAT3(signal transducer and activator of transcription 3) and cell cycle regulator p14 in a molecular pathological workout of the radical prostatectomy specimen).
early biochemical relapse | 5 years
  To evaluate, if the applied parameters of multiparametric metabolic imaging with FEC- and PSMA-PET/MRI are associated with the evidence of an early biochemical relapse after a PSA nadir <0.2ng/ml after primary treatment in a two years follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Imaging and Image-guided Therapy, Vienna, Austria

REFERENCES:
- [Derived] Ning J, Spielvogel CP, Haberl D, Trachtova K, Stoiber S, Rasul S, Bystry V, Wasinger G, Baltzer P, Gurnhofer E, Timelthaler G, Schlederer M, Papp L, Schachner H, Helbich T, Hartenbach M, Grubmuller B, Shariat SF, Hacker M, Haug A, Kenner L. A novel assessment of whole-mount Gleason grading in prostate cancer to identify candidates for radical prostatectomy: a machine learning-based multiomics study. Theranostics. 2024 Aug 1;14(12):4570-4581. doi: 10.7150/thno.96921. eCollection 2024. PMID 39239512
- [Derived] Papp L, Spielvogel CP, Grubmuller B, Grahovac M, Krajnc D, Ecsedi B, Sareshgi RAM, Mohamad D, Hamboeck M, Rausch I, Mitterhauser M, Wadsak W, Haug AR, Kenner L, Mazal P, Susani M, Hartenbach S, Baltzer P, Helbich TH, Kramer G, Shariat SF, Beyer T, Hartenbach M, Hacker M. Supervised machine learning enables non-invasive lesion characterization in primary prostate cancer with [68Ga]Ga-PSMA-11 PET/MRI. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1795-1805. doi: 10.1007/s00259-020-05140-y. Epub 2020 Dec 19. PMID 33341915
- [Derived] Aksoy O, Pencik J, Hartenbach M, Moazzami AA, Schlederer M, Balber T, Varady A, Philippe C, Baltzer PA, Mazumder B, Whitchurch JB, Roberts CJ, Haitel A, Herac M, Susani M, Mitterhauser M, Marculescu R, Stangl-Kremser J, Hassler MR, Kramer G, Shariat SF, Turner SD, Tichy B, Oppelt J, Pospisilova S, Hartenbach S, Tangermann S, Egger G, Neubauer HA, Moriggl R, Culig Z, Greiner G, Hoermann G, Hacker M, Heery DM, Merkel O, Kenner L. Thyroid and androgen receptor signaling are antagonized by mu-Crystallin in prostate cancer. Int J Cancer. 2021 Feb 1;148(3):731-747. doi: 10.1002/ijc.33332. Epub 2020 Oct 31. PMID 33034050